CLINICAL TRIAL: NCT06870890
Title: Impact of Sarcopenia on Dyspnea in Patients With Asthma
Acronym: MUDYSA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: AOI 2023 ROLLAND-DEBORD
Record Dates: First submitted 2025-02-24; First posted 2025-03-11 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Sarcopenia; Asthma; Dyspnea; Dyspnea; Asthmatic; Cytokines; Adipokines; Myokine; Muscle Disorder
Keywords: Asthma; Sarcopenia; Dyspnea
MeSH Terms: conditions — Sarcopenia; Asthma; Dyspnea; Muscular Diseases | interventions — Exercise Test; Surveys and Questionnaires; Restraint, Physical

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- All the patient included in the study (Experimental)
  Interventions: Diagnostic Test: muscle evaluation; Biological: Dosage; Diagnostic Test: Cardiopulmonary exercise test; Combination Product: Questionnaire and Physical Exam

INTERVENTIONS:
Diagnostic Test: muscle evaluation — The investigators will evaluate the muscle mass and muscle strenght for all patients included
Biological: Dosage — Evaluation of the cinetic of biomarkers during exercise
  Other Names: Others dosages at rest only; Dosage of biomarkers at rest and after exercise
Diagnostic Test: Cardiopulmonary exercise test — CPET
Combination Product: Questionnaire and Physical Exam — Evaluating dyspnea, anxiety, sleep, physical activity, quality of life

SUMMARY:
Dyspnea in asthma, is mainly due to airway obstruction but can be caused by several alternative diagnoses.

The impact of sarcopenia on dyspnea in patients with asthma is unknown. Sarcopenic asthma had a reduced physical activity and is associated with airway obstruction compared to non-sarcopenic asthma. In patients with obstructive pulmonary disease, sarcopenia is associated with shallow breathing and diverse sensory and affective components of exertional dyspnea .

The morbidity of sarcopenia is also increased by systemic inflammation and the production of inflammatory cytokines as found in inflammatory airway obstruction.

The investigators will investigate the prevalence and impact of sarcopenia in asthmatics patients. This will enable to better manage sarcopenia in asthmatic patients, understand its origins and personalize treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Patient affiliated to a social security scheme.
* Patient capable of giving free, informed, written and signed consent.
* Asthmatic patients with a diagnosis made by a pulmonologist on GINA level 4 or 5 treatment
* ACT asthma control score < 20
* Patient judged by the investigator to be able to to perform a maximal exercise test.

Exclusion Criteria:

* Patient under guardianship/trusteeship/supervision of justice
* Pregnant or breast-feeding women
* Unstable heart disease
* Patients who have been smoking or have stopped smoking for less than 5 years,

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-03-25 (Estimated); Primary Completion 2025-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Variation in the intensity of dyspnea during exercise mesured with Borg scale (0-10) according to the presence of sarcopenia | From baseline (at rest) to the end of the exercise
  Recording of Borg's dyspnea score during exercise on a scale of 0 (no dyspnea) to 10 (major dyspnea)

SECONDARY OUTCOMES:
Variation in exercise-induced release of biomarkers according to the presence of sarcopenia | at rest = baseline / right after the end of exercice / 45 minutes after the end of exercice
  Variation of cytokine as IL-1, IL-6, IL-8, IL-10 and TNF-alpha plasma concentrations (pg/mL) ; adipokines ; myokines
Difference in muscle mass (kg) on impedancemetry according to the presence of sarcopenia | Baseline
Difference on maximum aerobic capacity (VO2 max in L/mn) , according to the presence of sarcopenia | immediately after the exercise test
  Difference on physical activity
Difference in fat mass (kg) on impedancemetry according to the presence of sarcopenia | At baseline

CONTACTS AND LOCATIONS:
Overall Officials: Camille ROLLAND-DEBORD, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France

IPD SHARING:
Plan to Share IPD: No